CLINICAL TRIAL: NCT00510575
Title: Surgical Outcomes Using Variable Rod Diameters in the Treatment of Idiopathic Scoliosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Terri Green, Clinical Data Coordinator, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCLA-0123
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Scoliosis
Keywords: Juvenile Scoliosis; Adolescent Scoliosis; Scoliosis Management; Spinal Fusion; Scoliosis instrumentation; Juvenile or Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects in this arm will receive the 5.5mm stainless steel instrumentation rod.
  Interventions: Device: Spinal rod
- 2 (Active Comparator): Subjects in this arm will receive a 6.35mm stainless steel instrumentation rod.
  Interventions: Device: Spinal rod

INTERVENTIONS:
Device: Spinal rod — Posterior spinal fusion using a 5.5 or 6.35 size rod

SUMMARY:
There are two rod sizes routinely used for the correction of juvenile and adolescent idiopathic scoliosis, 5.5mm and 6.35mm, typically stainless steel. Currently there is no scientific evidence supporting the superiority of one size rod relative to the other. This study will evaluate the amount of radiographic correction obtained using the 5.5mm versus the 6.35mm spinal instrumentation rods.

DETAILED DESCRIPTION:
For the correction of Juvenile and Adolescent idiopathic scoliosis, companies offer and surgeons use varying rod sizes not based on scientific evidence, but because of personal preference, availability and company loyalty. To date there has been no literature evaluating the benefit or harm of one rod size versus the other. Our dual-arm prospective study will evaluate the amount of radiographic correction obtained using the 5.5mm versus the 6.35mm stainless steel instrumentation rods. These are both standard rods used in the community for this particular procedure, thus no additional risk exists for the patient. The results of this study will help guide surgeons in their decision making process when faced with the multitude of options offered by implant manufactures.

Comparison(s): 5.5mm stainless steel spinal rod versus 6.35mm stainless steel spinal rod for correction of juvenile and idiopathic scoliosis curves.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Juvenile or Adolescent Idiopathic Scoliosis
* Anticipated spinal fusion surgery

Exclusion Criteria:

* Individuals younger than 11 years and older than 18 years
* Individuals with scoliosis carrying additional diagnoses of illness.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Radiographic measurements of curve angles and balance. | Pre-operatively, 6 wks post-op, 1 & 2 year post-op.

SECONDARY OUTCOMES:
Scoliosis Research Society-30 (SRS-30) questionnaire | Pre-operatively, 6 wks post-op, 1 & 2 year post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Otsuka, MD, Study Director — Shriners Hospitals for Children - Los Angeles; Richard Bowen, MD, Principal Investigator — Shriners Hospitals for Children - Los Angeles
Locations (1):
- Shriners Hospitals for Children - Los Angeles, Los Angeles, California, United States